CLINICAL TRIAL: NCT06994442
Title: Optimizing Pain Treatment in Children On Mechanical Ventilation
Acronym: OPTICOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-12028276; U01HD116260 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation; Pediatric Acute Respiratory Failure; Analgesics, Opioid; Sedation and Analgesia
Keywords: Acetaminophen; Ketorolac; Non-opioids; Acute Respiratory Failure in Children; Mechanically Ventilated Children in the ICU; Pediatric Delirium; Pain Treatment; opioids; sedation
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intravenous Acetaminophen (IV-A) + Intravenous Placebo (Experimental): Participants receive intravenous acetaminophen and intravenous placebo every 6 hours, alongside open-label opioids per standard of care, for up to 5 days.
  Interventions: Drug: Acetaminophen; Drug: Placebo
- Intravenous Ketorolac (IV-K) + Intravenous Placebo (Experimental): Participants receive intravenous ketorolac and intravenous placebo every 6 hours, alongside open-label opioids per standard of care, for up to 5 days.
  Interventions: Drug: Ketorolac; Drug: Placebo
- Intravenous Acetaminophen (IV-A) + Intravenous Ketorolac (IV-K) (Experimental): Participants receive intravenous acetaminophen and intravenous ketorolac every 6 hours, alongside open-label opioids per standard of care, for up to 5 days.
  Interventions: Drug: Acetaminophen; Drug: Ketorolac
- Intravenous Placebo + Intravenous Placebo (Placebo Comparator): Participants receive intravenous placebo infusions every 6 hours, alongside open-label opioids per standard of care, for up to 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Intravenous (IV) dose, 15 mg/kg* (maximum 600 mg) every 6 h for 5 days.
  *Note: For children <28 days old, dose will be 12.5 mg/kg every 6 hours, as per U.S. Food and Drug Administration (FDA) recommendations. The dosing of acetaminophen for intravenous infusion will follow the current Acetaminophen for injection labeling based on the participant's age and weight.
  Arms: Intravenous Acetaminophen (IV-A) + Intravenous Ketorolac (IV-K); Intravenous Acetaminophen (IV-A) + Intravenous Placebo
Drug: Ketorolac — IV dose; 0.5mg/kg (maximum 30 mg) every 6 h for 5 days 4.1.d. *Note: Ketorolac for intravenous bolus administration is currently labeled for multiple-dose treatment in adults. For patients under 65 years of age, the recommended dose is 30 mg every 6 hours, with a maximum daily dose of 120 mg. For patients 65 years or older, renally impaired patients, and those weighting less than 50 kg, the recommended dose is 15 mg every 6 hours, with a maximum daily dose of 60 mg. In this study, we will be limiting ketorolac to <15 mg per dose, with a maximum of 60 mg per day.
  Arms: Intravenous Acetaminophen (IV-A) + Intravenous Ketorolac (IV-K); Intravenous Ketorolac (IV-K) + Intravenous Placebo
Drug: Placebo — Placebos will be normal saline solution, i.e., 0.9% NaCl. In order to maintain blinding, the investigational pharmacy will dispense placebo in a volume to match the corresponding study drug.
  Arms: Intravenous Acetaminophen (IV-A) + Intravenous Placebo; Intravenous Ketorolac (IV-K) + Intravenous Placebo; Intravenous Placebo + Intravenous Placebo

SUMMARY:
In this clinical trial, investigators want to learn more about using non-opioid pain medications for children with acute respiratory failure. Right now, doctors give these children opioids to help with pain while they are on the ventilator, but investigators don't know if this is the best way to manage their pain. Even with strong doses of opioids, more than 90% of these children still feel pain. Other pain medicines, like acetaminophen (also called Tylenol) and ketorolac (also called Toradol), are available but aren't commonly used because we don't know if they help. The goal of this clinical trial is to test if acetaminophen and/or ketorolac can improve pain control and reduce the need for stronger pain medications (opioids) in these children.

To learn more about this, participants will be randomly placed in one of four study treatment groups. This means that a computer will decide by chance which group each participant is in, not the doctors running the study. Each group will receive a combination of intravenous acetaminophen, ketorolac or a harmless substance called a placebo. In this clinical trial, placebos help investigators see if the actual medications (acetaminophen and ketorolac) work better than something that doesn't contain medicine. By comparing participants who get the real medicine with those who get the placebo, investigators can find out if these medications effectively decrease pain.

DETAILED DESCRIPTION:
The OPTICOM (Optimizing Pain Treatment In Children On Mechanical Ventilation) study is a multicenter, randomized, double-blind, placebo-controlled clinical trial designed to improve pain management and reduce opioid exposure in critically ill children requiring invasive mechanical ventilation (MV) for acute respiratory failure (ARF).

More than 24,000 children annually in the United States require MV for ARF, yet current analgesic management relies heavily on opioids, often resulting in suboptimal pain control and significant risks including physiological dependence, withdrawal, delirium, and prolonged hospitalization. Despite the high-dose opioid use, over 90% of these children experience inadequate pain relief. There are currently no evidence-based, pediatric-specific guidelines to optimize analgesia in this population.

OPTICOM will evaluate whether the administration of intravenous acetaminophen (IV-A) and/or intravenous ketorolac (IV-K), as non-opioid adjuncts, can reduce pain and opioid exposure in this vulnerable population. A total of approximately 644 participants aged 2 months to 17 years 6 months, requiring MV and opioid infusions, will be randomized in a 1:1:1:1 ratio into one of four treatment arms: (1) IV-A + placebo, (2) IV-K + placebo, (3) IV-A + IV-K, or (4) placebo + placebo. Study drugs will be administered for a maximum of 5 days. Opioid and benzodiazepine use will continue as open-label per local standard of care.

The study employs a factorial design with stratified randomization by site. The analysis plan includes multivariable Poisson regression models to evaluate the independent and combined effects of IV-A and IV-K on primary and secondary outcomes. Sample size calculations provide >90% power to detect meaningful differences in pain control and opioid reduction.

ELIGIBILITY:
Inclusion Criteria:

1. At least 2 months of age to 17 years 6 months; AND
2. Acute Respiratory Failure requiring endotracheal intubation; AND
3. Opioid infusion planned or started; AND
4. Expected duration of Invasive Mechanical Ventilation > 48 hours

Exclusion Criteria:

1. History of allergic-type reaction to either acetaminophen or non-steroidal anti-inflammatory (NSAID) medications; OR
2. Active peptic ulcer disease, recent gastrointestinal bleeding or perforation, or history of peptic ulcer disease or gastrointestinal bleeding; OR
3. Expected need for continuous neuromuscular blockade for more than 24 hours following intubation; OR
4. Requirement for tight temperature control (defined as the requirement for continuous administration of antipyretic medications to prevent secondary injuries associated with fever); OR
5. Platelet count < 100,000/microliter; OR
6. Known liver disease (defined as pre-existing diagnosis of hepatic insufficiency, or a serum ALT > 5 times upper limit of normal or serum total bilirubin > 2 times the upper limit of normal, as defined by hospital laboratory standards); OR
7. Known kidney disease (defined as pre-existing diagnosis of renal insufficiency, or an estimated creatinine clearance < 30 mL/min/m2 obtained within the previous 24-hours prior to eligibility, or high risk of renal failure due to volume depletion); OR
8. Current treatment with extracorporeal therapies (e.g., ECMO, CVVH, plasma exchange); OR
9. Cardiac bypass surgery within the past 24 hours prior to eligibility; OR
10. Requirement for the patient to receive lithium, pentoxifylline or probenecid as part of their routine care; OR
11. Unable to obtain consent and randomize within 12 hours of eligibility, OR
12. Positive pregnancy test; OR
13. Coma, Vegetative State, or Brain Death (Pediatric Cerebral Performance Category (PCPC) score of 5 or 6) suspected or confirmed; OR
14. Cardiac arrest has occurred within 72 hours of eligibility criteria being met; OR
15. Limitations in care in place at the time of eligibility, or anticipated to be considered during the 5-day study period, OR
16. Use of high dose NSAIDS within the prior 6 months, OR
17. Suspected or confirmed cerebrovascular bleeding or hemorrhagic diathesis

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 644 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Acute Pain Episodes | First 5 days of mechanical ventilation or until extubation, whichever comes first
  Pain will be assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) score. Coma will be defined using standardized sedation scales. The number of time periods where the participant is both pain-free (FLACC <4) and coma-free will be recorded.

SECONDARY OUTCOMES:
Opioid Exposure | First 5 days of mechanical ventilation or until extubation, whichever comes first
  Opioid exposure will be quantified in morphine milligram equivalents per kilogram during the first 5 days of mechanical ventilation.
Benzodiazepine Exposure | First 5 days of mechanical ventilation or until extubation, whichever comes first
  Total benzodiazepine exposure (in midazolam milligram equivalents per kilogram) during the first 5 days of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Chani Traube, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (15):
- United States (15):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Health/Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Wisconsin Children's, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including baseline, outcome, and adverse event data will be shared via NIH-approved repositories (e.g., HEAL KIDS Data Platform) within 12 months after publication of primary results. Access will be granted to qualified researchers with a methodologically sound proposal and appropriate agreements, for academic research, meta-analyses, and other approved studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will be available no later than 12 months after publication of the primary results and for at least 5 years thereafter.
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal. Researchers must agree to a data use agreement, and requests will be reviewed by the study team and the Data Coordinating Center.